CLINICAL TRIAL: NCT07186530
Title: HPV Self-Collection in Novel Settings to Increase Cervical Cancer Screening
Brief Title: Offering HPV Self-Collection in Novel Healthcare Settings to Improve Uptake of Cervical Cancer Screening
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 25-000735; NCI-2025-05848 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Cervical Carcinoma; Human Papillomavirus Infection; Human Papillomavirus-Related Cervical Carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms; Papillomavirus Infections | interventions — Practice Guidelines as Topic; Standard of Care; Electronic Health Records

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (HPV self-collection) (Experimental): Participants receive a portal message inviting them to schedule and complete cervical cancer screening via HPV self-collection at an Express Care clinic. Participants are also informed they can choose the usual care of a cervical cancer screening test with their primary care team in clinic instead. Participants who complete screening receive standard follow-up care.
  Interventions: Other: Best Practice; Other: Communication Intervention; Other: Electronic Health Record Review; Procedure: HPV Self-Collection; Procedure: Standard Follow-Up Care
- Arm II (usual care) (Active Comparator): Participants receive usual care and standard follow-up care on study.
  Interventions: Other: Best Practice; Other: Electronic Health Record Review; Procedure: Standard Follow-Up Care

INTERVENTIONS:
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
Other: Communication Intervention — Receive portal message
  Arms: Arm I (HPV self-collection)
Other: Electronic Health Record Review — EHR reviewed to assess whether recommended follow-up was completed, if follow-up was indicated.
  Other Names: Electronic Health Record (EHR) Review; EHR Review
Procedure: HPV Self-Collection — Complete HPV self-collection
  Other Names: HPV Self Collection; Human Papillomavirus Self-Collection; HPV Self-Collection in a healthcare setting
  Arms: Arm I (HPV self-collection)
Procedure: Standard Follow-Up Care — Receive standard follow-up care

SUMMARY:
This clinical trial evaluates whether offering human papillomavirus (HPV) self-collection for cervical cancer screening at Mayo Clinic Express Care clinics improves uptake of cervical cancer screening and receipt of appropriate follow-up care. Cervical cancer is preventable through vaccination, screening, and treatment of pre-cancerous conditions. However, cervical cancer screening rates have declined over the past 25 years, and an estimated 25% of women are unscreened or overdue for screening. Usual care at Mayo Clinic currently includes annual portal or letter communications in the form of scheduled outreach to request scheduling an appointment for cervical cancer screening, as well as reminders from clinicians during clinic appointments. Cervical cancer screening at Mayo Clinic is most often done with a pelvic speculum exam with cervical swabs collected in the office by a clinician. HPV self-collection is Food and Drug Administration-approved and already used in clinical practice, but offering this method of screening in the novel setting of Express Care clinics that have expanded nighttime and weekend hours may improve rates of cervical cancer screening and receipt of appropriate follow-up care.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 30-63 years old receiving primary care with a provider at Mayo Clinic in Rochester and who self-identify as asymptomatic (i.e., no pelvic pain, abnormal vaginal bleeding or abnormal vaginal discharge)
* Qualify for average risk cervical cancer screening per United States Preventive Services Task Force (USPSTF) guidelines but are overdue by >= 1 year, including those who have never been screened
* Must have an active Patient Online Services account (patient portal), approval for research contact status in portal/Epic and documentation of Minnesota (MN) research authorization, and health insurance coverage

Exclusion Criteria:

* History of hysterectomy
* Cervical cancer
* Cervical intraepithelial neoplasia (CIN) 2-3
* In utero diethylstilbestrol (DES) exposure
* HIV+
* Use of chronic immunosuppressant medication
* Known to be pregnant
* Medicare-covered women are NOT eligible as Medicare does not cover primary HPV testing by clinician-collection or self-collection [related to outdated Centers for Medicare & Medicaid Services (CMS) cervical cancer screening coverage rules for Medicare that date back to 2015, 3 years before primary HPV screening was endorsed by USPSTF]

Ages: 30 Years to 63 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2030-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Cervical cancer screening test | Up to 6 months from trial enrollment
  Assessed by the number of participants who complete cervical cancer screening collection from invitation to complete a self-collected vaginal swab for HPV testing at Mayo Clinic Express Care clinics compared to the number of participants who complete screening with a clinician-collected cervical swab or self-collected vaginal swab at a primary care office.

SECONDARY OUTCOMES:
Follow-up of abnormal results | Up to 6 months from date of test
  Assessed by the number of participants who complete follow-up for abnormal results obtained by self-collection or clinician-collection.

CONTACTS AND LOCATIONS:
Overall Officials: Kathy L. Maclaughlin, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials